CLINICAL TRIAL: NCT06285045
Title: Randomized Controlled Study on Roujin Formula in the Treatment of Fibromyalgia Syndrome With Blood Deficiency and Liver Depression
Brief Title: Study on Roujin Formula in the Treatment of Fibromyalgia Syndrome With Blood Deficiency and Liver Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Juan Jiao, chief physician, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2060302-1703-05
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Fibromyalgia Syndrome
Keywords: Fibromyalgia syndrome; Blood deficiency and liver depression；; Roujin Formula; Clinical trial
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Roujin Formula group (Experimental): Roujin Formula : angelica, bupleurum, radix paeoniae alba, etc. Medication method : oral 1 bag ( 150ml ) each time, 2 times a day. Treatment course : 8 weeks.
  Interventions: Drug: Roujin Formula
- Control group (No Intervention): Placebo : According to the internationally accepted standard, one-tenth of the dose of Roujin Formula was used to prepare a placebo, which was similar to Roujin Formula in appearance, color, taste or smell, and packaging. Medication method : oral 1 bag ( 150ml ) each time, 2 times a day. Treatment course : 8 weeks.

INTERVENTIONS:
Drug: Roujin Formula — 48 eligible participants with FMS of blood deficiency and liver depression syndrome were selected and randomly divided into treatment group(n=24)and control group(n=24). The treatment group was given Roujin Foumula 150mL,twice a day; The control group was given Roujin Foumula placebo 150mL,twice a day,the study period was 8 weeks. The evaluation points were 0 weeks,4 weeks,and 8 weeks of treatment,and follow-up to 12 weeks. To evaluate the effect changes before and after treatment,FIQR score、VAS score、PSQI score、BDI score and SF-36 PCS、MCS score were used as secondary efficacy evaluation indexes. SPSS23.0 was used to analyze the data.
  Arms: Roujin Formula group

SUMMARY:
To evaluate the efficacy and safety of Roujin Formula in the treatment of fibromyalgia syndrome(FMS)patients with blood deficiency and liver depression through a randomized,single-blind,placebo-parallel controlled exploratory clinical trial study,and to provide reliable clinical evidence for the treatment of fibromyalgia syndrome with Roujin Formula. 48 eligible participants with FMS of blood deficiency and liver depression syndrome were selected and randomly divided into treatment group(n=24)and control group(n=24). The treatment group was given Roujin Foumula 150mL,twice a day; The control group was given Roujin Foumula placebo 150mL,twice a day,the study period was 8 weeks. The evaluation points were 0 weeks,4 weeks,and 8 weeks of treatment,and follow-up to 12 weeks. To evaluate the effect changes before and after treatment,FIQR score、VAS score、PSQI score、BDI score and SF-36 PCS、MCS score were used as secondary efficacy evaluation indexes. SPSS23.0 was used to analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* 1. Meet the 1990 American College of Rheumatology (ACR) Research Classification Criteria for filbromyalgia;
* 2. Be over 18 years of age;
* 3. Sign informed consent.

Exclusion Criteria:

* 1.patients with rheumatoid arthritis, systemic lupus erythematosus, dermatomyositis, ankylosing spondylitis and other rheumatic diseases ;
* 2.severe liver and kidney dysfunction;
* 3.severe cardiovascular and cerebrovascular diseases and other diseases ;
* 4.pregnant or lactating women ;
* 5.had taken drugs for the treatment of this disease in the last 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
The change of the revised Fibromyalgia Impact Questionnaire (FIQR) from baseline | baseline,4 weeks, 8 weeks, 12 weeks
  A self-administered questionnaire with 10 subscales, measuring fibromyalgia symptoms and function domains. FIQR total score ranges from 0 to 100, with higher scores indicating more severe symptoms.
The change of the Visual Analogue Scale (VAS) for pain from baseline | baseline,4 weeks, 8 weeks, 12 weeks
  Pain VAS, range, 0 to 10 cm, where higher scores indicated the perceived pain to be more severe.

SECONDARY OUTCOMES:
The change of the Pittsburgh Sleep Quality Index(PSQI) from baseline | baseline,4 weeks, 8 weeks, 12 weeks
  Scores on the Pittsburgh Sleep Quality Index (PSQI) range from 0 to 21, with higher scores indicating worse sleep quality.
The change of the Beck depression inventory(BDI) from baseline | baseline,4 weeks, 8 weeks, 12 weeks
  The Beck II Depression Inventory (BDI) assesses the severity of depressive symptoms. Scores range from 0 to 39, with higher scores indicate a greater degree of depression severity.
The change of the Short Form-36 Health Status Questionnaire(SF-36) from baseline | baseline,4 weeks, 8 weeks, 12 weeks
  The Short Form-36 Health Status Questionnaire (SF-36), which measured health-related quality of life (range, 0 to 100, with higher scores indicating better perceived health status).The Short Form-36 Health Status Questionnaire (SF-36), which measured health-related quality of life (range, 0 to 100, with higher scores indicating better perceived health status).

CONTACTS AND LOCATIONS:
Locations (1):
- Juan Jiao, Beijing, Beijing Municipality, China